CLINICAL TRIAL: NCT00895596
Title: A PhaseII, Open-Label, Multinational, Multi-Centre, Sequential Group, Dose-Escalation Study to Assess the Safety and Antiviral Activity of LB80380 for 12 Weeks in Patients With Lamivudine-Refractory Chronic Hepatitis B
Brief Title: Safety and Efficacy Study of LB80380 in the Patients With Lamivudine-Refractory Chronic Hepatitis B
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: LG Life Sciences, Ltd.
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: BVCL004
Record Dates: First submitted 2009-05-07; First posted 2009-05-08 (Estimated); Last update posted 2009-05-08 (Estimated); Status verified 2009-05

CONDITIONS: Chronic Hepatitis B
Keywords: Chronic hepatitis B; Lamivudine resistant; YMDD mutant type
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — ((1-((2-amino-9H-purin-9-yl)methyl)cyclopropyl)oxy)methylphosphonic acid dipivoxyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- LB80380 30mg (Experimental): LB80380 30mg
  Interventions: Drug: LB80380
- LB80380 60mg (Experimental): LB80380 60mg
  Interventions: Drug: LB80380
- LB80380 90mg, (Experimental): LB80380 90mg
  Interventions: Drug: LB80380
- LB80380 150mg (Experimental): LB80380 150mg
  Interventions: Drug: LB80380
- LB80380 240mg (Experimental): LB80380 240mg
  Interventions: Drug: LB80380

INTERVENTIONS:
Drug: LB80380 — Total treatment period: 12 weeks, followed by 24 weeks of treatment with adefovir dipivoxil 10mg

SUMMARY:
The purpose of the study is to investigate the safety and the antiviral activity of ascending multiple oral doses of LB80380 for 12 weeks in adults with lamivudine-refractory chronic hepatitis B infection.

DETAILED DESCRIPTION:
LB80380, an oral prodrug, is a promising candidate nucleoside analogue with antiviral activity against wild-type HBV. LB80380 is undergoing clinical development by LG Life Sciences for use in the treatment of chronic HBV infection and for treatment of lamivudine-resistant disease.

In this study, the treatment period was divided into two parts: a 4-week treatment period with dose escalation assessment (Part 1), followed by an 8-week extension period (Part 2).

During Part 1, patients received LB80380 and LVD 100 mg once daily for 4 weeks. Each patient was then given only LB80380 for an additional 8 weeks (Part 2) unless dose-limiting toxicity (DLT) was observed during Part 1. At each dose level, all patients were to complete at least Part 1 of the treatment period before enrolment into the next Dose Group could commence. Dose escalation to the next group was not to be initiated if more than two patients experienced DLT during Part 1 in the previous Dose Group. Additionally, patients enrolled in LB80380 150mg and 240mg groups who agreed to participate in the pharmacokinetic (PK) analyses visited the study site the day before Week 12 for blood sampling. Follow-up period was 24 weeks, and patients were treated with adefovir dipivoxil during the follow-up period. During the study, patients were evaluated for changes from baseline in serum HBV DNA. Safety was evaluated on the basis of occurrence of AEs and changes from baseline in clinical laboratory parameters, physical examination findings, and vital signs.

ELIGIBILITY:
Inclusion Criteria:

* Compensated chronic hepatitis B patient
* Presence of serum HBsAg for more than 6 months.
* Presence of HBeAg for more than 1 month with compensated liver disease
* Confirmation of YMDD mutants (M552V, M552I and its related double mutant at L528M) by genotyping of the YMDD motif using line probe assay (INNO-LiPA HBV DR assay)
* Screening HBV DNA value higher than or equal to 1,000,000 copies/mL (measured by the COBAS Amplicor HBV Monitor™ assay)
* Screening ALT value between 1.5 and 10 x ULN

Exclusion Criteria:

* Co-infection with hepatitis C or D virus (HCV or HDV) or HIV
* Pregnancy or breast-feeding
* Previous treatment with nucleoside analogue or any other treatment for HBV except for lamivudine within 6 months prior to study entry
* Treatment with immunomodulatory agent or corticosteroids within 6 months prior to study entry.
* De-compensated liver disease
* Screening alpha-fetoprotein (AFP) value > 20 ng/mL, and a follow-up ultrasonography performed prior to baseline shows findings indicative of HCC.
* Presence of anti-HBs at screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2004-03; Primary Completion 2006-08 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Mean serum HBV DNA level (log10) reduction from the baseline at Week 12 | Week 12

SECONDARY OUTCOMES:
Proportion of patients with HBeAg seroconversion at 12 weeks Proportion of patients with HBsAg seroconversion at 12 weeks Proportion of patients with ALT normalization at 12 weeks Safety assessment during the whole study period | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Lung Lai, Dr, Principal Investigator — Queen Mary Hospital, Hong Kong
Locations (4):
- Queen Mary Hospital, Hong Kong, China
- South Korea (3):
  - Korea University Medical Center, Seoul
  - Severance Hospital of Yonsei University, Seoul
  - The Catholic University of Korea, Kangnam St. Mary's Hospital, Seoul

REFERENCES:
- [Derived] Yuen MF, Han KH, Um SH, Yoon SK, Kim HR, Kim J, Kim CR, Lai CL. Antiviral activity and safety of LB80380 in hepatitis B e antigen-positive chronic hepatitis B patients with lamivudine-resistant disease. Hepatology. 2010 Mar;51(3):767-76. doi: 10.1002/hep.23462. PMID 20091678